CLINICAL TRIAL: NCT02829710
Title: Implementation and Evaluation of a Paediatric Nurse-driven Sedation Protocol in a Paediatric Intensive Care Unit
Brief Title: Implementation and Evaluation of a Pediatric Nurse-driven Sedation Protocol in a PICU
Acronym: SEDATIDE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0312
Record Dates: First submitted 2016-06-28; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Analgesia; Deep Sedation
Keywords: Analgesia; intensive care units; clinical protocol; deep sedation; nursing assessment
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group 1 : pre implementation group: All children aged less than 18 years, requiring mechanical ventilation for at least 24 hours and admitted in PICU between January 2013 and December 2013.
  Prior to implementation of the protocol, analgesia and sedation were managed by the attending physician's order.
- group 2 : post implementation group: All children aged less than 18 years, requiring mechanical ventilation for at least 24 hours and admitted in PICU between May 2014 and March 2015.
  Nurses managed analgesia and sedation following an algorithm, including COMFORT-B scale.
  Interventions: Behavioral: Nurse-driven sedation protocol

INTERVENTIONS:
Behavioral: Nurse-driven sedation protocol — The nurse-driven sedation protocol included the COMFORT-B scale. Initial doses were chosen by the physicians then all changes were made by the nurses with the aim of attaining an optimal range of analgesia and sedation, which was defined as values from 11 to 17 on the COMFORT-B score.
  Groups: group 2 : post implementation group

SUMMARY:
Management of analgesia and sedation is an integral component of the medical care of a critically-ill child. Its role is to assure comfort and safety to a patient undergoing painful cares and technical procedures; it can also be, in particular situations like acute respiratory distress syndrome or acute brain injury, a full processing treatment.

Sedation involves, most of the time, the association of an opioid and a sedative. The use of these drugs is difficult in children, because of a specific metabolism, inducing tolerance and withdrawal in case of prolonged administration.

The COMFORT-BEHAVIOR (COMFORT-B) scale is a validated, simple, reliable and reproducible score evaluating sedation and analgesia. Sedation scoring systems must be used regularly to avoid inadequate sedation.

Excessive sedation is associated with poor outcomes like prolonged mechanical ventilation, longer hospitalisation and more frequent withdrawal symptoms. Adult and paediatric data suggest that goal-directed sedation algorithms allow a more appropriate adaptation of the treatment to the patient's need and permit a reduction in the duration of mechanical ventilation.

The objective was to evaluate the impact of a nurse-driven sedation protocol in a paediatric intensive care unit on duration of mechanical ventilation, total doses and duration of medications, Paediatric Intensive Care Unit (PICU) length of stay, incidence of ventilator-associated-pneumonia and occurrence of withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically-ventilated patients aged from 0 to 18 years receiving sedation for more than 24 hours

Exclusion Criteria:

* Patients with tracheostomy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children aged from 0 to 18 years, requiring mechanical ventilation for at least 24 hours admitted in a PICU between January 2013 and December 2013 and between May 2014 and March 2015.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation (days) | Over the PICU stay of each child (Day 5)

SECONDARY OUTCOMES:
Total doses of sedatives (unit/kg) | Over the PICU stay of each child (Day 5)
Occurrence of withdrawal symptoms | Over the PICU stay of each child (Day 5)
Length of PICU stay (days) | Over the PICU stay of each child (Day 5)

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Bordet, MD, Principal Investigator — service de réanimation pédiatrique, Hôpital Femme Mère Enfant (HFME), Hospices Civils de Lyon
Locations (1):
- service de réanimation pédiatrique, Hôpital Femme Mère Enfant (HFME), Hospices Civils de Lyon, 59 Boulevard Pinel, Bron, France